CLINICAL TRIAL: NCT00459940
Title: "Can Growth Hormone's Lipolytic and Insulin-Antagonistic Effects be Modified by Peroxisome Proliferator-Activated Gamma Agonists?"
Brief Title: The Effects of TZD on Fat Metabolism and Insulin Sensitivity in GH-Replaced GHD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20030288
Record Dates: First submitted 2007-04-12; First posted 2007-04-13 (Estimated); Last update posted 2007-04-13 (Estimated); Status verified 2007-04

CONDITIONS: Growth Hormone Deficiency
Keywords: Growth hormone; Lipolysis; Insulin resistance; Pioglitazone; Growth hormone replaced growth hormone deficient adults
MeSH Terms: conditions — Dwarfism, Pituitary; Insulin Resistance | interventions — Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Pioglitazone

SUMMARY:
In the present double blind, placebo-controlled, parallel study we evaluated the impact of 12 weeks thiazolidinedione (TZD) administration on basal and insulin-stimulated substrate metabolism in growth hormone-replaced adults with growth hormone deficiency.

DETAILED DESCRIPTION:
In human subjects GH (Growth Hormone) acutely antagonises the effects of insulin on glucose uptake in skeletal muscle and increases the hepatic glucose production of humans. This has clinical implications for patients with active acromegaly, in whom the prevalence of glucose intolerance and overt diabetes mellitus is increased. It is also of significance in relation to GH replacement therapy in GH-deficient adults not least when considering that a substantial proportion of these patients are insulin resistant in the GH-untreated state. There is evidence to indicate that the acute insulin antagonistic effects may be balanced with time by the favourable effects of GH on body composition and physical fitness, but the data are ambiguous. The mechanism underlying these effects of GH are not fully characterised, but there is experimental evidence of a causal linked to the concomitant stimulation of lipolysis, since GH-induced insulin resistance is partly abrogated when lipolysis is pharmacologically suppressed. This is noteworthy since elevated levels of free fatty acids (FFA) are also implicated in the pathogenesis of insulin resistance in patients with the metabolic syndrome and type 2 diabetes mellitus. Thiazolidinediones (TZDs) are insulin sensitizers which function as highaffinity agonists for the nuclear peroxisome-proliferator-activated receptor (PPAR) gamma, which improve insulin sensitivity in T2DM. PPAR gamma is a nuclear receptor expressed mainly in adipocytes, which activates the transcription of genes involved in lipid and glucose metabolism. Administration of TZD in T2DM enhances insulin-stimulated glucose uptake via mechanisms including a lowering of circulating FFA and a redistribution of fat away from hepatocytes and myocytes and into peripheral adipocytes. To our knowledge, the impact of TZDs on GH-induced insulin resistance has not previously been reported. Experimental data in human subjects on this issue are of potential importance not only in relation to patients with abnormal GH status, but also regarding our understanding of the pathogenesis of insulin resistance in general and the complex actions of PPAR gamma activation in particular.

ELIGIBILITY:
Inclusion Criteria:

* Growth hormone replaced (minimum 6 months) growth hormone deficient men
* Age over 18 years

Exclusion Criteria:

* Ischemic coronary disease, defined by EF<0.6, former myocardial infarction, angina pectoris or actual treatment of cardiac insufficiency
* Actual or former malignancy, except intracranial neoplasia that caused the participants pituitary disease, provided that there was clinical evidence for permanent remission
* Blood donation within 6 months
* Excessive alcohol consumption
* Known allergic reaction from contents of test drug
* Radioactive radiation exposure in terms of treatment or study enrollment within one year
* Liver insufficiency
* Insulin treatment

Ages: 19 Years to 71 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2004-09; Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Circulating FFA level
FFA turnover
Lipid oxidation

CONTACTS AND LOCATIONS:
Overall Officials: Jens OL Jorgensen, MD, Principal Investigator — University of Aarhus
Locations (1):
- Medical Department M, The Medical Research Laboratories, Aarhus University Hospital, Aarhus C, Denmark

REFERENCES:
- [Background] Boden G, Cheung P, Mozzoli M, Fried SK. Effect of thiazolidinediones on glucose and fatty acid metabolism in patients with type 2 diabetes. Metabolism. 2003 Jun;52(6):753-9. doi: 10.1016/s0026-0495(03)00055-6. PMID 12800103
- [Background] Racette SB, Davis AO, McGill JB, Klein S. Thiazolidinediones enhance insulin-mediated suppression of fatty acid flux in type 2 diabetes mellitus. Metabolism. 2002 Feb;51(2):169-74. doi: 10.1053/meta.2002.29981. PMID 11833043
- [Background] Alford FP, Hew FL, Christopher MC, Rantzau C. Insulin sensitivity in growth hormone (GH)-deficient adults and effect of GH replacement therapy. J Endocrinol Invest. 1999;22(5 Suppl):28-32. PMID 10442567
- [Background] Spiegelman BM. PPAR-gamma: adipogenic regulator and thiazolidinedione receptor. Diabetes. 1998 Apr;47(4):507-14. doi: 10.2337/diabetes.47.4.507. PMID 9568680
- [Background] Nielsen S, Moller N, Christiansen JS, Jorgensen JO. Pharmacological antilipolysis restores insulin sensitivity during growth hormone exposure. Diabetes. 2001 Oct;50(10):2301-8. doi: 10.2337/diabetes.50.10.2301. PMID 11574412
- [Background] Nielsen S, Moller N, Pedersen SB, Christiansen JS, Jorgensen JO. The effect of long-term pharmacological antilipolysis on substrate metabolism in growth hormone (GH)-substituted GH-deficient adults. J Clin Endocrinol Metab. 2002 Jul;87(7):3274-8. doi: 10.1210/jcem.87.7.8597. PMID 12107236
- [Background] Norrelund H, Djurhuus C, Jorgensen JO, Nielsen S, Nair KS, Schmitz O, Christiansen JS, Moller N. Effects of GH on urea, glucose and lipid metabolism, and insulin sensitivity during fasting in GH-deficient patients. Am J Physiol Endocrinol Metab. 2003 Oct;285(4):E737-43. doi: 10.1152/ajpendo.00092.2003. Epub 2003 Jun 10. PMID 12799313